CLINICAL TRIAL: NCT03292081
Title: Comparison Between Optical Frequency Domain Imaging and Intravascular Ultrasound in Percutaneous Coronary Intervention Guidance for Biolimus A9 Eluting Stent Implantation
Brief Title: Comparison Between OFDI and IVUS in PCI Guidance for Biolimus A9 Eluting Stent Implantation
Acronym: MISTIC-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fujita Health University (Other)
Responsible Party: Principal Investigator, Yukio Ozaki, Professor, Department of Cardiology, Fujita Health University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-106
Record Dates: First submitted 2017-08-29; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease
Keywords: Intracoronary Imaging; Optical Frequency Domain Imaging; Intravascular Ultrasound; Percutaneous Coronary Intervention; Drug Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFDI-guided PCI (Experimental)
  Interventions: Device: OFDI
- IVUS-guided PCI (Active Comparator)
  Interventions: Device: IVUS

INTERVENTIONS:
Device: OFDI — PCI under OFDI guidance
  Other Names: LUNAWAVE imaging console; Fastview imaging catheter
  Arms: OFDI-guided PCI
Device: IVUS — PCI under IVUS guidance
  Other Names: VISIWAVE imaging console; ViewIT imaging catheter
  Arms: IVUS-guided PCI

SUMMARY:
The aim of this study is to assess clinical safety and efficacy of percutaneous coronary intervention (PCI) using a newer generation drug-eluting stent (DES) in the context of optical frequency domain imaging (OFDI) guidance or intravascular ultrasound (IVUS) guidance.

DETAILED DESCRIPTION:
Intracoronary imaging techniques provide clinically useful information in the setting of PCI, such as lesion severity, tissue characterization, vessel sizing, and stent optimization. Current evidences suggest potential advantage of intracoronary imaging guidance in reducing the risk of major adverse cardiac events after stent implantation over conventional PCI under angiographic guidance alone. IVUS has been clinically used in two decades and it is known as one of the most dominant intracoronary imaging technique. OFDI is a new light-based intracoronary imaging technology which provides higher image resolution and higher-speed pullback compared to those of IVUS. Given the different properties between ultrasound-based IVUS and light-based OFDI, treatment and clinical impact of these two imaging techniques would be different.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable coronary artery disease who have symptoms or myocardial ischemia proven by non-invasive or invasive stress test.

Exclusion Criteria:

* Renal insufficiency with estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m2
* Left ventricular ejection fraction (LVEF) <30% or history of congestive heart failure
* Acute coronary syndrome within 7 days after onset
* Considered as inappropriate for drug-eluting stent (DES) use or dual antiplatelet therapy for one year after the index procedure
* Life expectancy within one year
* Lesion length estimated by quantitative coronary angiography (QCA) >28mm
* Chronic total occlusion
* Left main stem lesion
* Bifurcation requiring side branch balloon dilatation
* Severely calcified lesion
* Other conditions by which physicians in charge judged inappropriate to enroll the patients because of safety concern.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2014-06-12 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2017-10-25 (Estimated)

PRIMARY OUTCOMES:
Minimum lumen area assessed by OFDI | 8 months

SECONDARY OUTCOMES:
Cardiovascular mortality | 8 months
Target vessel myocardial infarction | 8 months
Target lesion revascularization | 8 months
Apposition of stent struts assessed by OFDI | 8 months
Tissue coverage of stent struts assessed by OFDI | 8 months
Quantitative Coronary Angiography (QCA) | 8 months

OTHER OUTCOMES:
Integrated Backscatter IVUS (IB-IVUS) | 0 month (pre-procedure)
  Plaque components including lipid pool, fibrosis, dense fibrosis or calcification
Detectable external elastic lamina (EEL) arc assessed by OFDI | 0 month (pre-procedure)

CONTACTS AND LOCATIONS:
Locations (1):
- Fujita Health University, Toyoake, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Muramatsu T, Ozaki Y, Nanasato M, Ishikawa M, Nagasaka R, Ohota M, Hashimoto Y, Yoshiki Y, Takatsu H, Ito K, Kamiya H, Yoshida Y, Murohara T, Izawa H; MISTIC-1 Investigators. Comparison Between Optical Frequency Domain Imaging and Intravascular Ultrasound for Percutaneous Coronary Intervention Guidance in Biolimus A9-Eluting Stent Implantation: A Randomized MISTIC-1 Non-Inferiority Trial. Circ Cardiovasc Interv. 2020 Nov;13(11):e009314. doi: 10.1161/CIRCINTERVENTIONS.120.009314. Epub 2020 Oct 27. PMID 33106049